CLINICAL TRIAL: NCT06272630
Title: A Multicenter, Randomized, Placebo Controlled, Double-blinded, Phase 4 Study to Evaluate the Efficacy and Safety of DWJ1464 in Patients with Chronic Liver Disease
Brief Title: Study to Evaluate the Efficacy and Safety of DWJ1464 in Patients with Chronic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWJ1464401
Record Dates: First submitted 2023-04-06; First posted 2024-02-22 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DWJ1464 (Experimental): UCDA 100 mg, TID
  Interventions: Drug: DWJ1464
- Placebo of DWJ1464 (Placebo Comparator): Placebo of DWJ1464, TID
  Interventions: Drug: Placebo of DWJ1464

INTERVENTIONS:
Drug: DWJ1464 — DWJ1464, TID, Duration of administration: 8 weeks, Visit: every 4 week
  Arms: DWJ1464
Drug: Placebo of DWJ1464 — Placebo of DWJ1464, TID, Duration of administration: 8 weeks, Visit: every 4 week
  Arms: Placebo of DWJ1464

SUMMARY:
This study aims to assess the effect of DWJ1464 on improvement of liver function in patients with Chronic liver disease. Patients with Chronic liver disease aged 19 years or over will participate in the study. The study design is a multi-center double-blinded randomized placebo-controlled trial. The patients were diagnosed with Chronic liver disease based on our criteria and were randomized to either the placebo or DWJ1464 administration group. Primary endpoint was the change of ALT level after 8 weeks compared to the baseline. Secondary endpoints included the change of ALT level after 4 weeks, the change rate of ALT level after 8 weeks and improvement of fatigue, compared to the baseline. the adverse effect of DWJ1464 were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic liver disease(presented with abnormal serum ALT levels >6 months and twice continuously or abnormal area of liver through medical imaging test within 6 months
* Abnormal serum ALT levels at screening and baseline

Exclusion Criteria:

* Subjects who have diseases that liver cirrhosis, liver cancer, renal dysfunction etc.
* Subjects who are taking medications or supplements related to chronic liver disease, fatigue.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
At 8 weeks, the change of ALT level compared to baseline | 8 weeks after randomization

SECONDARY OUTCOMES:
At 4 weeks, the change of ALT level compared to baseline | 4 weeks after randomization
At 4, 8 weeks, the change of AST level compared to baseline | 4, 8 weeks after randomization
At 4, 8 weeks, the change of liver function comparator GGT level compared to baseline | 4, 8 weeks after randomization
At 8 weeks, the change of liver function comparator Fibrotest compared to baseline | 4, 8 weeks after randomization
At 8 weeks, the change of liver function comparator Fibroscan compared to baseline | 4, 8 weeks after randomization
At 4, 8 weeks, the change of K-CFQ(Korean version of Chalder Fatigue Scale) scores, compared to the baseline | 4, 8 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jae Young Jang, MD, PhD, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- SoonChunHyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided